CLINICAL TRIAL: NCT01386892
Title: Immunological Characterization of Blood of Normal Individuals
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2011H0007
Record Dates: First submitted 2011-04-27; First posted 2011-07-01 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Heathly Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Saliva Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteer: Healthy Volunteer without lung disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention for this study

SUMMARY:
This study seeks to obtain normal samples of blood, saliva and urine to serve as controls for other approved protocols and for analysis. These include determination of the functional capabilities of cells, proteins, nucleic acids and microvesicles obtained from peripheral blood including plasma, serum and cellular fraction from normal individuals. Saliva and urine will have similar testing which may also be compared to the blood testing results. The ongoing objective varies from investigation to investigation but in general the investigational goals are to better understand the immune function of normal volunteers and compare it to immune function in disease states.

DETAILED DESCRIPTION:
Blood will be obtained via peripheral venipuncture. The blood will be divided into components (e.g. plasma, serum, microvesicles, and cells) then analyzed. Flow cytometry will be used to determine cell and microvesicle subsets. RNA will be extracted from the various components of blood and will be subjected to gene and microRNA profiling to determine gene expression. DNA will be isolated from the cells to be used in studies investigating epigenetic regulation of genes identified in the screens. Protein will also be isolated from the multiple components to examine the impact of genetic regulation by epigenetic mechanisms or microRNA on protein expression. Peripheral blood mononuclear cells will be placed in tissue culture for study.

Saliva and urine will be obtained the same day as blood for testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no chronic or acute illnesses, or taking medication which in the opinion of the PI would impact the analyses being conducted.
* At least 18 years or older.
* Are capable of reading, understanding and providing written informed consent.

Exclusion Criteria:

* Non-English speaking.
* Individuals under 18 years old.
* Woman who believe they are or may be pregnant. (Based on self reporting. Pregnancy testing will not be conducted for the purposes of this study)
* Individuals experiencing acute or chronic illnesses which in the opinion of the PI would impact the analyses being conducted.
* Currently taking prescription or over the counter medication which in the opinion of the PI would impact the analyses being conducted.
* Individual has donated blood more than twice in the last week or the amount to be drawn will exceed the maximum allowance in the last 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants may also be recruited by word of mouth or via public advertising. This study is open to all eligibile healthy adult volunteers regardless of gender, age and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2015-01-05 (Actual); Study Completion 2015-01-05 (Actual)

PRIMARY OUTCOMES:
Blood content differences between the lung disease and healthy control populations | Day 1
  Test for differences in the blood of individuals with lung disease and normal healthy controls.

SECONDARY OUTCOMES:
Genetic expression of relevant genes between the lung disease and healthy control populations | Day 1
  Test for genetic differences in the blood of individuals with lung disease and normal healthy controls.
Saliva and urine analysis results compared to blood content results between the lung disease and healthy control populations. | Day 1
  Analyze saliva and urine along with the blood sample in order to compare the information in the blood with the saliva and urine.
Identify diagnostic and prognostic indicators for lung disease | December 2020
  Develop and test possible diagnostic and prognostic indicators for various lung diseases.
Develop possible treatment for lung disease | December 2020
  Develop and test possible reprogramming of blood cells to promote vessel formation as a way to prevent tumor metastases and modify the progression of specific lung diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Clay Marsh, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States